CLINICAL TRIAL: NCT00316719
Title: Phase III Study of Adefovir Dipivoxil Tablets in Patients With Compensated Chronic Hepatitis B -Comparative Study Against Lamivudine-
Brief Title: Adefovir Dipivoxil In Compensated Chronic Hepatitis B Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADF105220
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Results first posted 2009-08-03 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Chronic Hepatitis B
Keywords: treatment naive; CHB; adefovir; monotherapy
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Lamivudine; adefovir dipivoxil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Adefovir Dipivoxil (ADV) (Experimental)
  Interventions: Drug: ADV group
- Lamivudine (LAM) (Active Comparator)
  Interventions: Drug: LAM group

INTERVENTIONS:
Drug: LAM group — Subjects took one LAM 100mg tablet orally once daily and one ADV placebo tablet orally once daily.
  Other Names: Lamivudine
  Arms: Lamivudine (LAM)
Drug: ADV group — Subjects took one ADV 10mg tablet orally once daily and one LAM placebo tablet orally once daily.
  Other Names: adefovir dipivoxil
  Arms: Adefovir Dipivoxil (ADV)

SUMMARY:
This study is designed to compare the efficacy and safety of adefovir dipivoxil 10 mg with lamivudine 100 mg in Japanese patients with compensated chronic hepatitis B over 52-week periods.

ELIGIBILITY:
Inclusion criteria:

* Have compensated chronic hepatitis B.
* Have not been treated with anti HBV agents with antiproliferative activity against. However, previous Interferon (IFN) therapy is permitted.
* Ability to read, understand, and sign the informed consent.
* Have a positive serum HBV-DNA >= 1,000,000 copies/mL and ALT level 50-500 U/L

Exclusion criteria:

* Having or suspected of having liver cancer.
* Co-infected with Hepatitis C virus (HCV) or Human Immunodeficiency virus (HIV).
* Autoimmune hepatitis.
* Received any previous transplantation or having a plan for any transplantation.
* Existence of any serious complication, except hepatitis B.

Ages: 16 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2006-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Groups:
- Adefovir (ADV): ADV 10 mg orally once daily for 52 weeks
- Lamivudine (LAM): LAM 100 mg orally once daily for 52 weeks
Period: Overall Study
Arm/Group | Adefovir (ADV) | Lamivudine (LAM)
Started | 52 | 53
Completed | 50 | 47
Not Completed | 2 | 6
Not completed — Adverse Event | 0 | 6
Not completed — Consent withdrawn | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adefovir (ADV) | Lamivudine (LAM) | Total
Number analyzed (Participants) | 50 | 52 | 102
Age Continuous [Mean (Standard Deviation); unit: years] | 44 (9.73) | 43.9 (9.95) | 44 (9.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 17 | 26
  Male | 41 | 35 | 76
Race/Ethnicity, Customized [Number; unit: Number of participants]
  Asian | 50 | 52 | 102
Region of Enrollment [Number; unit: participants]
  Japan | 50 | 52 | 102

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Hepatitis B Virus (HBV) DNA at Week 52
Description: Change from baseline was the difference of the HBV DNA copy numbers (log10) in serum collected by blood draw between baseline and Week 52
Time Frame: Baseline and Week 52
Population: Per Protocol Set (PPS): participants in the Full Analysis Set (all subjects who entered the study, received at least one dose of investigational product, and had at least one efficacy assessment after the treatment initiation) population with no major protocol violations
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Adefovir (ADV) | Lamivudine (LAM)
Number analyzed (Participants) | 50 | 52
log10 copies/mL | -3.69 (1.169) | -3.40 (1.896)
Statistical Analysis 1: Comparison: Adefovir (ADV) vs Lamivudine (LAM); Test type: Non-Inferiority or Equivalence — This is a Non-inferiority Analysis with the margin of -1.0; p < 0.001, ANCOVA; Mean Difference (Net) = -0.33, 95% CI [-0.94 to 0.28], Standard Error of Mean 0.309

2. Secondary Outcome: Percentage of Participants With HBV DNA Loss (<400 Copies/mL) at Week 52
Description: The percentages of participants with an HBV DNA level in serum of less than 400 copies/mL, which is the lower limit of detection (HBV DNA loss) at Week 52
Time Frame: Week 52
Population: PPS
Measure: Number; unit: Percentage of participants
Arm/Group | Adefovir (ADV) | Lamivudine (LAM)
Number analyzed (Participants) | 50 | 52
Percentage of participants
  <400 copies/mL | 46.0 | 50.0
  >400 copies/mL | 54.0 | 50.0

3. Secondary Outcome: Time to Onset of HBV DNA Loss (< 400 Copies/mL)
Description: Time to onset of an HBV DNA level in serum of less than 400 copies/mL was summarized using the Kaplan-Meier method. Regarding the Measured Values, the median time to onset and its upper limit for the ADV group and the upper limit of the median time to onset for the LAM group are non-estimable because they are not observed until the end of the study. The lower limit of the median time to onset for the ADV and LAM groups are 36.0 and 20.0, respectively. The median time to onset for the LAM group is 28.0
Time Frame: From Baseline to Week 52
Reporting Status: Not Posted
Measure: Median (95% Confidence Interval); unit: weeks

4. Secondary Outcome: Percentage of Participants With Hepatitis B e Antigen (HBeAg) Loss at Week 52
Description: Participants with loss of Hepatitis B e antigen (HBeAg) in serum collected by blood draw: Cheminoluminescent Immuno Assay (CLIA) method
Time Frame: Week 52
Population: PPS: participants who were positive for HBeAg at baseline
Measure: Number; unit: percentage of participants
Arm/Group | Adefovir (ADV) | Lamivudine (LAM)
Number analyzed (Participants) | 36 | 37
percentage of participants
  With loss of HBeAg | 16.7 | 16.2
  Positive for HBeAg | 93.3 | 93.8

5. Secondary Outcome: Percentage of Participants With Hepatitis B e Antigen/Antibody (HBeAg/Ab) Seroconversion at Week 52
Description: Participants with loss of Hepatitis B e antigen (HBeAg) and positive for anti-Hepatitis B e antibody (HBeAb) in serum collected by blood draw: CLIA method
Time Frame: Week 52
Population: PPS: participants who were positive for HBeAg and negative for HBeAb at baseline
Measure: Number; unit: Percentage of participants
Arm/Group | Adefovir (ADV) | Lamivudine (LAM)
Number analyzed (Participants) | 31 | 34
Percentage of participants
  With HBeAg/Ab seroconversion | 9.7 | 5.9
  Without HBeAg/Ab seroconversion | 90.3 | 94.1

6. Secondary Outcome: Time to Onset of HBeAg Loss
Description: Time to onset with loss of HBeAg in serum collected by blood draw was summarized using the Kaplan-Meier method.: CLIA method. Regarding the Measured Values, the median time to onset and its lower limit and its upper limit for all groups are non-estimable because they are not observed until the end of the study.
Time Frame: From Baseline to Week 52
Reporting Status: Not Posted
Measure: Median (95% Confidence Interval); unit: weeks

7. Secondary Outcome: Time to Onset of HBeAg/Ab Seroconversion
Description: Time to onset of HBeAg/Ab seroconversion in serum collected by blood draw was summarized using the Kaplan-Meier method.: CLIA method. Regarding the Measured Values, the median time to onset and its lower limit and its upper limit for all groups are non-estimable because they are not observed until the end of the study.
Time Frame: From Baseline to Week 52
Reporting Status: Not Posted
Measure: Median (95% Confidence Interval); unit: weeks

8. Secondary Outcome: Percentage of Participants With Hepatitis B s Antigen (HBsAg) Loss at Week 52
Description: Participants with loss of Hepatitis B s antigen (HBsAg) in serum collected by blood draw: CLIA method
Time Frame: Week 52
Population: PPS: participants who were positive for HBsAg at baseline
Measure: Number; unit: percentage of participants
Arm/Group | Adefovir (ADV) | Lamivudine (LAM)
Number analyzed (Participants) | 50 | 52
percentage of participants
  With loss of HBsAg | 0.0 | 0.0
  Positive for HBsAg | 100.0 | 100.0

9. Secondary Outcome: Percentage of Participants With Hepatitis B s Antigen/ Antibody (HBsAg/Ab) Seroconversion at Week 52
Description: Participants with loss of Hepatitis B s antigen (HBsAg) and positive for anti-Hepatitis B s antibody (HBsAb) in serum collected by blood draw: CLIA method
Time Frame: Week 52
Population: PPS: participants who were positive for HBsAg and negative for HBsAb at baseline
Measure: Number; unit: percentage of participants
Arm/Group | Adefovir (ADV) | Lamivudine (LAM)
Number analyzed (Participants) | 46 | 45
percentage of participants
  With HBsAg/Ab seroconversion | 0.0 | 0.0
  Without HBsAg/Ab seroconversion | 100.0 | 100.0

10. Secondary Outcome: Mean Alanine Aminotransferase (ALT) Level at Week 52
Description: Summary statistics were displayed for serum ALT.
Time Frame: Week 52
Population: PPS
Measure: Mean (Standard Deviation); unit: Units per Liter
Arm/Group | Adefovir (ADV) | Lamivudine (LAM)
Number analyzed (Participants) | 50 | 47
Units per Liter | 32.3 (14.72) | 33.0 (28.12)

11. Secondary Outcome: Percentage of Participants With Alanine Aminotransferase (ALT) Normalization at Week 52
Description: ALT normalization was defined as an ALT value that was in the normal range (<= 45IU/L; upper limit of normal [ULN]) at Week 52 of the participants whose ALT values were abnormal (>45IU/L) at baseline
Time Frame: Week 52
Population: PPS: Participants with an abnormal ALT value (>ULN) at baseline
Measure: Number; unit: Percentage of participants
Arm/Group | Adefovir (ADV) | Lamivudine (LAM)
Number analyzed (Participants) | 46 | 51
Percentage of participants
  With ALT normalization | 82.6 | 78.4
  Without ALT normalization | 17.4 | 21.6

12. Secondary Outcome: Time to Onset of ALT Normalization
Description: Time to onset of ALT normalization was summarized using the Kaplan-Meier method.
Time Frame: From Baseline to Week 52
Population: PPS: Participants with abnormal ALT value (>ULN) at baseline
Measure: Median (95% Confidence Interval); unit: Week 52
Arm/Group | Adefovir (ADV) | Lamivudine (LAM)
Number analyzed (Participants) | 46 | 51
Week 52 | 12.0 [8.0 to 16.0] | 12.0 [12.0 to 16.0]

13. Secondary Outcome: Rate of Emergence of Resistant Virus at Week 52
Description: Participants with resistant mutation at Week 52. LAM resistant mutation (enzyme-linked mini-sequencing assay): rtM204I/V; ADV resistant mutation (direct sequencing assay): rtN236T or rtA181T/V in HBV DNA ; rt: reverse transcriptase gene
Time Frame: Week 52
Population: PPS
Measure: Number; unit: Percentage of participants
Arm/Group | Adefovir (ADV) | Lamivudine (LAM)
Number analyzed (Participants) | 50 | 52
Percentage of participants
  With resistant mutation | 0 | 28.8
  Without resistant mutation | 100 | 71.2

ADVERSE EVENTS:
Arm/Group | Adefovir (ADV) | Lamivudine (LAM)
Serious Adverse Events (participants affected / at risk) | 0/52 | 4/53
Other Adverse Events (participants affected / at risk) | 39/52 | 47/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adefovir (ADV) (N=52) | Lamivudine (LAM) (N=53)
Hepatitis (Hepatobiliary disorders) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adefovir (ADV) (N=52) | Lamivudine (LAM) (N=53)
Diarrhea (Gastrointestinal disorders) | 7 | 6
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 1 | 4
Vomiting (Gastrointestinal disorders) | 0 | 3
Nasopharyngitis (Infections and infestations) | 11 | 19
Upper respiratory tract inflammation (Infections and infestations) | 7 | 10
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Eczema (Skin and subcutaneous tissue disorders) | 5 | 3
Blood creatine phosphokinase increased (Investigations) | 5 | 4
Malaise (General disorders) | 2 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Headache (Nervous system disorders) | 1 | 4
Hepatitis (Hepatobiliary disorders) | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.